CLINICAL TRIAL: NCT03158727
Title: A Phase Ib/IIa, Randomised, Double Blind, Parallel Group, Placebo Controlled, Multicentre Study to Assess the Safety and Efficacy of Expanded Cx611 Allogeneic Adipose-derived Stem Cells (eASCs) for the Intravenous Treatment of Adult Patients With Severe Community-acquired Bacterial Pneumonia and Admitted to the Intensive Care Unit
Brief Title: Cx611-0204 SEPCELL Study
Acronym: SEPCELL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Collaborators: European Commission (Other); Centre Hospital Regional Universitaire de Limoges (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Hospital San Carlos, Madrid (Other)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cx611-0204; 2015-002994-39 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-18 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Bacterial Pneumonia
Keywords: Biologic Therapy
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cx611 (Experimental): Subjects treated in an intensive care unit for sCABP, but that may be screened at the emergency department, will receive SoC therapy according to local guidelines plus two intravenous central line infusions of Cx611 at a fixed dose of 160 million expanded allogeneic adipose-derived stem cells (eASCs) each.
  Interventions: Biological: Cx611
- Placebo (Placebo Comparator): Subjects treated in an intensive care unit for sCABP, but that may be screened at the emergency department, will receive SoC therapy according to local guidelines plus two intravenous central line infusions of Ringer Lactate.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Cx611 — Two intravenous infusions, one on day 1 and another one on day 3.
  Arms: Cx611
Other: Placebo — Two intravenous infusions, one on day 1 and another one on day 3.
  Arms: Placebo

SUMMARY:
The purpose of this randomised, multicentre, double-blind, placebo-controlled, phase Ib/IIa study is to assess the safety, tolerability and efficacy of eASCs (Cx611) administered intravenously as adjunctive therapy, therefore in addition to standard of care (SoC) therapy, to patients with severe community-acquired bacterial pneumonia (sCABP).

The completion of this study will contribute to the basic knowledge on stem cells and their mode-of-action, and has a large translational character, i.e. to document the safety and explore the efficacy of Cx611 in patients with sCABP.

DETAILED DESCRIPTION:
The purpose of this randomised, multicentre, double-blind, placebo-controlled, phase Ib/IIa study is to assess the safety, tolerability and efficacy of eASCs (Cx611) administered intravenously as adjunctive therapy, therefore in addition to standard of care (SoC) therapy, to patients with severe community-acquired bacterial pneumonia (sCABP).

The key objectives of this study are to:

Primary objective:

Investigate the safety profile of two allogeneic Cx611 80 mL infusions administered through a central line within 3 days (on days 1 and 3) at a dose of 160 million cells each (320 million cells total) and to monitor any adverse event and potential immunological host responses against the administered cells during 90 days of follow-up after the first infusion.

Secondary objective:

Explore the clinical efficacy of Cx611 in terms of a reduction of the duration of mechanical ventilation and/or need for vasopressors and/or improved survival, and/or clinical cure of the sCABP, and other efficacy-related endpoints.

ELIGIBILITY:
Inclusion criteria

1. Adult subjects of either gender (aged ≥18 years and ≤80 years old.)
2. Body weight between 50 kg and 100 kg.
3. Clinical diagnosis of acute (developed within ≤21 past days) community acquired bacterial pneumonia based on the presence of two relevant signs (fever, tachypnoea, leukocytosis, or hypoxemia) and radiographic findings of new pulmonary infiltrate/s.
4. Subjects with pneumonia of sufficient severity requiring ICU management and with at least one of the two following major criteria of severity present for less than 18 hours:

   1. Requiring invasive mechanical ventilation for respiratory failure due to pneumonia, or
   2. Requiring treatment with vasopressors (i.e., dopamine >5 mcg/kg/min or any dose of epinephrine, norepinephrine, phenylephrine or vasopressin) for at least 2 hours to maintain or attempt to maintain systolic blood pressure (SBP) >90 mm Hg (or mean arterial pressure [MAP] >70 mm Hg) after adequate fluid resuscitation (i.e. for shock).

   NOTE: Patients that are for 18 hours or more under high flow nasal cannula (HFNC) at ≥50 liters per minute and FiO2 ≥0.6 or under non-mechanical ventilation (NMV) are not eligible for the study
5. Female subject of no childbearing potential i.e. non-fertile, pre-menarche, permanently sterile (i.e. underwent hysterectomy, bilateral salpingectomy or bilateral ovariectomy) or post-menopausal (history of no menses for at least 12 months without an alternative medical cause) or Woman of childbearing potential* with a negative serum or urine pregnancy test (sensitive to 25 IU human chorionic gonadotropin [hCG]) and agree to use an adequate method of contraception for three months after the last dose of the IMP according to her preferred and usual life style. Adequate methods of female contraception for this study are: sexual abstinence (refraining from heterosexual intercourse), hormonal contraception (both progesterone-only or combined oestrogen and progesterone; both with inhibition of ovulation or where inhibition of ovulation is not the primary mechanism of action), intra-uterine device, bilateral tubal occlusion, condom use by male sexual partner(s) or medically-assessed successfully vasectomized male sexual partner(s).

   *A woman of childbearing potential is a woman between menarche and post-menopause (history of no menses for at least 12 months without an alternative medical cause) unless she has undergone hysterectomy, bilateral salpingectomy or bilateral ovariectomy Male subject agreeing to use one of the following methods of birth control according to his preferred and usual life style for three months after the last dose of the IMP: sexual abstinence (refraining from heterosexual intercourse), use of condoms or medically-assessed successful vasectomy , or having a female sexual partner(s) who is using an adequate method of contraception as described above.
6. Signed informed consent provided by the participant, the relatives or the designated legal representative according to local guidelines.

Exclusion criteria A patient will not be included in the study if he/she meets ANY of the following criteria:

1. Subjects with Hospital acquired (HAP)-, Health Care acquired (HCAP)- or Ventilator associated-pneumonia (VAP).
2. Subjects with pneumonia exclusively of viral or fungal origin*. Subjects with bacterial pneumonia co-infected with viruses and/or other microorganisms may be entered into the study.

   *Due to the short time window (up to 18 hours) between fulfillment of severity criteria (i.e. initiation of invasive mechanical ventilation or vasopressors administration, whichever comes first) and the start of the first dose of study treatment, patients with a pneumonia of suspected bacterial origin by any established standard diagnostic method routinely applied at the study site (e.g. urinary antigen test, rt-PCR) can be entered into the study (confirmation of bacterial origin must be obtained afterwards).
3. Subjects with known or suspected Pneumocystis jirovecii (formerly known as Pneumocystis carinii) pneumonia.
4. Subjects with an aspiration pneumonia.
5. Subjects with known active tuberculosis.
6. Subjects with a history of post-obstructive pneumonia.
7. Subjects with cystic fibrosis.
8. Subjects with any chronic lung disease requiring oxygen therapy at home.
9. Presence of infection in another organ location caused by same pathogen (e.g. pneumococcal meningitis in the context of pneumococcal pneumonia).
10. Subjects expected to have rapidly fatal disease within 72 hours after randomisation.
11. Inability to maintain a mean arterial pressure ≥50 mmHg prior to screening despite the presence of vasopressors and intravenous fluids.
12. Subjects not expected to survive for 3 months due to other pre-existing medical conditions such as end-stage neoplasm or other diseases.
13. Subjects with a history of malignancy in the 5 years prior to screening, except for successfully surgically treated non-melanoma skin malignancies.
14. Subjects with known primary immunodeficiency disorder or with HIV infection and acquired immune deficiency syndrome (AIDS) with CD4 count <200 cells/mm^3 or not receiving highly active antiretroviral therapy (HAART) for HIV.
15. Subjects receiving immunosuppressant therapy (including chronic treatment with anti-tumour necrosis factor alpha (TNFα ) or on chronic high doses of steroids (single administration of ≥2 mg/kg body weight or 20 mg/day of prednisone or equivalent for ≥2 weeks).
16. Chronic granulocytopenia, not thought to be due to sepsis, as evidenced by an absolute neutrophil count <500 per µL>21 days prior to onset of pneumonia symptoms.
17. Subjects who received stem cell therapy, or allogenic transplantation (organ or bone marrow transplant) within the past 6 months.
18. Subjects receiving treatment with a biological agent (e.g. antibodies, cells), immunotherapy or plasma exchange treatment within the last 8 weeks.
19. Subjects currently receiving, or having received another investigational medication within 90 days prior to start of the study (or 5 half-lives of the investigational compound, whichever is longer).
20. Known allergies or hypersensitivity to Penicillin or Streptomycin and/or any component of CryoStor® CS10.
21. Subjects with a known liver function impairment associated with liver cirrhosis (Child Pugh C) or known oesophageal varices.
22. Subjects hospitalised within the previous 15 days.
23. Conditions resulting in a New York Heart Association or Canadian Cardiovascular Society Class IV functional status.
24. End-stage neuromuscular disorders (e.g. motor neuron diseases, myasthenia gravis, etc.) or cerebral disorders that impair weaning.
25. Patients with quadriplegia (traumatic or otherwise).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- Belgium (4):
  - Clinique Universitaire Saint-Luc, Brussels, Brussels Capital
  - UZ Brussel, Brussels
  - CHU Sart Tilman, Liège
  - Clinique Saint-Pierre, Ottignies
- France (12):
  - Centre Hospitalier d'Angoulême, Angoulême
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - CHU Bocage, Dijon
  - Centre Hospitalier Departemental les Ouidairies, La Roche-sur-Yon
  - Centre Hospitalier Départemental les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Limoges - CHU Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Regional d'Orleans, Orléans
  - CHRU de Strasbourg, Strasbourg
  - CHU TOURS - Hôpital Bretonneau, Tours
- Azienda Ospedaliera San'Andrea. UOC Anestesia e Terapia Intensiva, Roma, Italy
- Klaipėda Republican Hospital, The Pulmonology and Allergology Department, Klaipėda, Lithuania
- St. Olavs Hospital, Department of Intensive care Clinical Immunology and Infectious Disease, Trondheim, Norway
- Spain (14):
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic I Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Laterre PF, Sanchez Garcia M, van der Poll T, Wittebole X, Martinez-Sagasti F, Hernandez G, Ferrer R, Caballero J, Cadogan KA, Sullivan A, Zhang B, de la Rosa O, Lombardo E, Francois B; SEPCELL Study Group. The safety and efficacy of stem cells for the treatment of severe community-acquired bacterial pneumonia: A randomized clinical trial. J Crit Care. 2024 Feb;79:154446. doi: 10.1016/j.jcrc.2023.154446. Epub 2023 Oct 31. PMID 37918129
- [Derived] Laterre PF, Sanchez-Garcia M, van der Poll T, de la Rosa O, Cadogan KA, Lombardo E, Francois B. A phase Ib/IIa, randomised, double-blind, multicentre trial to assess the safety and efficacy of expanded Cx611 allogeneic adipose-derived stem cells (eASCs) for the treatment of patients with community-acquired bacterial pneumonia admitted to the intensive care unit. BMC Pulm Med. 2020 Nov 25;20(1):309. doi: 10.1186/s12890-020-01324-2. PMID 33238991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in Belgium, France, Lithuania, and Spain from 30 Jan 2017 to 07 July 2020.
Pre-assignment Details: Adult participants with severe community-acquired bacterial pneumonia (sCABP) and admitted to the intensive care unit (ICU) were enrolled in 1 of the 2 treatment groups to receive Cx611 or placebo on Days 1 and 3.
Groups:
- Placebo: Participants received SoC therapy followed by two 80 mL central line infusions of placebo, intravenously, on Days 1 and 3.
- Cx611 160 mL: Participants received SoC therapy followed by two 80 mL central line infusions of Cx611, intravenously, on Days 1 and 3 at a fixed dose of 160 million eASCs (320 million cells total).
Period: Overall Study
Arm/Group | Placebo | Cx611 160 mL
Started | 42 | 42
Enrolled, Not Treated | 1 | 0
Completed | 25 | 23
Not Completed | 17 | 19
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Death | 11 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant doesn't want to come back to the hospital for the visit | 2 | 0
Not completed — Visit 11 not done by mistake | 0 | 1
Not completed — Enrolled, not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cx611 160 mL | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.43) | 61.1 (11.24) | 62.3 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 26 | 28 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 31 | 28 | 59
  Asian/Oriental | 1 | 0 | 1
  Hispanic | 1 | 1 | 2
  Latino | 2 | 1 | 3
  Unknown | 6 | 12 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 12 | 7 | 19
  Spain | 23 | 22 | 45
  Lithuania | 0 | 1 | 1
  France | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Day 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 37 | 40

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESIs are predefined adverse events (AEs) that required close monitoring and prompt reporting to the sponsor. Protocol-specific AEs considered as AESI for this study are thromboembolic events and hypersensitivity reactions such as anaphylaxis.
Time Frame: Baseline up to Day 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 9 | 7

3. Primary Outcome: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity reactions included anaphylaxis (changes in systolic and diastolic blood pressure, core temperature, respiratory rate [non-ventilated participants], heart rate), episodes of skin reactions and signs and symptoms of respiratory distress, which require therapeutic intervention including drugs and/or changes in mechanical ventilation setting. Number of participants with hypersensitivity reactions were reported for this outcome measure.
Time Frame: Baseline up to Day 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 1 | 0

4. Primary Outcome: Number of Participants With Markedly Abnormal Values of 12-lead Electrocardiogram (ECG) Parameters on Day 1
Time Frame: Day 1
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 3 | 7

5. Primary Outcome: Number of Participants With Markedly Abnormal Values of 12-lead Electrocardiogram (ECG) Parameters on Day 3
Time Frame: Day 3
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 5 | 4

6. Primary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Time Frame: Baseline up to Day 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 0 | 0

7. Primary Outcome: Number of Participants With Anti-human Leukocyte Antigen Complex (Anti-HLA)/Donor Antibodies At Day 1, 14, and 90
Time Frame: At Days 1, 14, and 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment. Here "number analyzed" are the participants who were evaluable for this outcome measure at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants
  Participants with Anti-HLA/Donor Antibodies at Day 1: number analyzed (Participants) | 37 | 40
  Participants with Anti-HLA/Donor Antibodies at Day 1 | 6 | 4
  Participants with Anti-HLA/Donor Antibodies at Day 14: number analyzed (Participants) | 36 | 32
  Participants with Anti-HLA/Donor Antibodies at Day 14 | 4 | 5
  Participants with Anti-HLA/Donor Antibodies at Day 90: number analyzed (Participants) | 28 | 21
  Participants with Anti-HLA/Donor Antibodies at Day 90 | 4 | 4

8. Secondary Outcome: Mechanical Ventilation and Vasopressors Treatment-free Days
Description: Participants with sCABP suffer either a respiratory failure that requires invasive mechanical ventilation and/or a severe hypotension that requires vasopressors. Number of days when participants were alive and free from mechanical ventilation and vasopressors were reported.
Time Frame: Baseline up to Day 28
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 19.0 [0 to 27] | 13.5 [0 to 25]

9. Secondary Outcome: Percentage of Participants Alive and Free of Both Mechanical Ventilation and Vasopressors at Day 29
Description: Participants with sCABP suffer either a respiratory failure that requires invasive mechanical ventilation and/or a severe hypotension that requires vasopressors. Percentage of participants who were alive and free of both mechanical ventilation and vasopressors at Day 29 were reported.
Time Frame: Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
percentage of participants | 78.0 | 64.3

10. Secondary Outcome: Percentage of Participants Alive and Free of Mechanical Ventilation at Day 29
Time Frame: Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
percentage of participants | 78.0 | 66.7

11. Secondary Outcome: Number of Ventilator Free Days (VeFD)
Description: VeFD are defined as one point for each day during the measurement period that participants are both alive and free from mechanical ventilation.
Time Frame: Baseline up to Day 28
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 19.0 [0 to 28] | 14.0 [0 to 28]

12. Secondary Outcome: Percentage of Participants Alive and Free of Vasopressors at Day 29
Time Frame: Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
percentage of participants | 85.4 | 76.2

13. Secondary Outcome: Number of Vasopressor Treatment-free Days (VaFD)
Description: VaFD over 28 days defined as one point for each day during the measurement period that participants are both alive and free of vasopressors.
Time Frame: Baseline up to Day 28
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 24.0 [0 to 28] | 23.5 [0 to 28]

14. Secondary Outcome: Time to End of Invasive Mechanical Ventilation
Description: Time in days, from the start date of invasive mechanical ventilation to the first stop date of invasive mechanical ventilation (that is, first time the participant ends mechanical ventilation), or death. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment. Here, "overall number of participants analyzed" are those who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 33 | 39
days | 7.7 [4.6 to 11.5] | 8.3 [4.6 to 12.4]

15. Secondary Outcome: Time to End of Invasive and/or Non-invasive Mechanical Ventilation
Description: Time in days, from the start date of invasive or non-invasive mechanical ventilation to the first stop date of invasive or non-invasive mechanical ventilation (that is, first time the participant ends mechanical ventilation), or death. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 29
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 33 | 39
days | 6.3 [3.3 to 10.3] | 4.7 [2.9 to 8.3]

16. Secondary Outcome: Time to End of Vasopressors Treatment
Description: Time in days, from the start date of vasopressors treatment to the first stop date of vasopressors treatment (that is, first time the participant ends vasopressors treatment), or death. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 29
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 33 | 34
days | 2.1 [1.4 to 3.0] | 2.0 [1.0 to 2.4]

17. Secondary Outcome: Number of Participants With sCABP Clinical Response Visit at Days 8-10, 14, and 29
Description: Cure:complete pneumonia resolution at baseline(BL),no new pneumonia symptoms/complications attributable.Non-response:failure related/unrelated to pneumonia:persistence/progression of BL signs/symptoms of pneumonia;BL radiographic abnormalities after atleast 2 days of treatment;development of new pulmonary/extra pulmonary findings consistent with active infection/development of new pulmonary infection/extrapulmonary infection requiring antimicrobial therapy;persistence/progression of BL signs/symptoms of severe sepsis;development of new signs/symptoms of severe sepsis;death due to sepsis.Non-response-failure unrelated to pneumonia:any cause of clinical response failure that in investigator's judgement is unrelated to index pneumonia(e.g.myocardial infarction, pulmonary thromboembolism, sepsis of urinary origin etc).Indeterminate:extenuating circumstances precluding classification to one of the above.
Time Frame: Days 8 to 10, 14, and 29
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants
  Days 8 to 10 (Cure): number analyzed (Participants) | 38 | 36
  Days 8 to 10 (Cure) | 18 | 21
  Days 8 to 10 (Failure not resulting in death): number analyzed (Participants) | 38 | 36
  Days 8 to 10 (Failure not resulting in death) | 8 | 6
  Days 8 to 10 (Indeterminate): number analyzed (Participants) | 38 | 36
  Days 8 to 10 (Indeterminate) | 11 | 9
  Days 8 to 10 (Missing): number analyzed (Participants) | 38 | 36
  Days 8 to 10 (Missing) | 1 | 0
  Day 14 (Cure): number analyzed (Participants) | 36 | 33
  Day 14 (Cure) | 24 | 24
  Day 14 (Failure not resulting in death): number analyzed (Participants) | 36 | 33
  Day 14 (Failure not resulting in death) | 5 | 4
  Day 14 (Indeterminate): number analyzed (Participants) | 36 | 33
  Day 14 (Indeterminate) | 6 | 4
  Day 14 (Missing): number analyzed (Participants) | 36 | 33
  Day 14 (Missing) | 1 | 1
  Day 29 (Cure): number analyzed (Participants) | 32 | 30
  Day 29 (Cure) | 30 | 26
  Day 29 (Failure not resulting in death): number analyzed (Participants) | 32 | 30
  Day 29 (Failure not resulting in death) | 1 | 1
  Day 29 (Indeterminate): number analyzed (Participants) | 32 | 30
  Day 29 (Indeterminate) | 0 | 3
  Day 29 (Missing): number analyzed (Participants) | 32 | 30
  Day 29 (Missing) | 1 | 0

18. Secondary Outcome: Time to sCABP Clinical Cure
Description: Cure is defined as complete resolution of pneumonia signs and symptoms present at baseline, no new symptoms or complications attributable to the pneumonia. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 13.0 [10.0 to 16.0] | 9.5 [8.0 to 14.0]

19. Secondary Outcome: Duration of Antibiotic Treatment
Time Frame: Baseline up to Day 29
Population: as for outcome 14
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 39 | 38
days | 9.0 [2 to 29] | 8.0 [1 to 29]

20. Secondary Outcome: Percentage of Participants With Pneumonia Recurrence or Reinfection After Clinical Cure
Description: Pneumonia recurrence is defined as a new acute clinical episode of pneumonia, after clinical cure of the episode that qualified the participant for the study, based on the presence of two relevant signs (fever, tachypnoea, leukocytosis, or hypoxemia) and radiographic findings of new pulmonary infiltrate/s or clinically significant worsening of previous ones. If a bacterial pathogen isolated in the recurrent episode is phenotypically different from the one isolated in the previous episode this will be considered as reinfection.
Time Frame: Days 14, 29, and 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment. Here, "overall number of participants analyzed" are those who were evaluable for this outcome measure. Here, "number analyzed" are the participants who were evaluable for the outcome measure at given time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 36 | 33
percentage of participants
  Day 14: Recurrence | 5.6 | 0
  Day 14: Reinfection | 8.3 | 6.1
  Day 29: Recurrence: number analyzed (Participants) | 32 | 30
  Day 29: Recurrence | 0 | 3.3
  Day 29: Reinfection: number analyzed (Participants) | 32 | 30
  Day 29: Reinfection | 0 | 0
  Day 90: Recurrence: number analyzed (Participants) | 28 | 25
  Day 90: Recurrence | 0 | 0
  Day 90: Reinfection: number analyzed (Participants) | 28 | 25
  Day 90: Reinfection | 0 | 0

21. Secondary Outcome: Time to Recurrence or Reinfection of Pneumonia After Clinical Cure at sCABP Clinical Response Assessments
Description: Pneumonia recurrence is defined as a new acute clinical episode of pneumonia, after clinical cure of the episode that qualified the participant for the study, based on the presence of two relevant signs (fever, tachypnoea, leukocytosis, or hypoxemia) and radiographic findings of new pulmonary infiltrates or clinically significant worsening of previous ones. If a bacterial pathogen isolated in the recurrent episode is phenotypically different from the one isolated in the previous episode this will be considered as reinfection. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 90
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 34 | 32
days | NA [NA to NA] — Median and 95% confidence interval could not be calculated because an insufficient number of participants had an event. | NA [NA to NA] — Median and 95% confidence interval could not be calculated because an insufficient number of participants had an event.

22. Secondary Outcome: 28-day All-cause Mortality
Time Frame: Day 28
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 6 | 8

23. Secondary Outcome: 28-day sCABP-associated Mortality
Time Frame: Day 28
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 0 | 1

24. Secondary Outcome: Survival at Baseline, Days 10, 20, 30, 40, 50, 60, 70, 80, and 90
Description: Survival data for percentage of participants at Baseline and at Days 10, 20, 30, 40, 50, 60, 70, 80, and 90 was assessed and reported.
Time Frame: At Baseline, Days 10, 20, 30, 40, 50, 60, 70, 80, and 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
percentage of participants
  Baseline | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Day 10 | 95.1 [81.9 to 98.8] | 88.1 [73.7 to 94.9]
  Day 20 | 87.5 [72.6 to 94.6] | 80.7 [65.0 to 89.8]
  Day 30 | 85.0 [69.5 to 93.0] | 80.7 [65.0 to 89.8]
  Day 40 | 77.0 [60.4 to 87.3] | 80.7 [65.0 to 89.8]
  Day 50 | 77.0 [60.4 to 87.3] | 75.3 [58.9 to 85.9]
  Day 60 | 77.0 [60.4 to 87.3] | 75.3 [58.9 to 85.9]
  Day 70 | 77.0 [60.4 to 87.3] | 75.3 [58.9 to 85.9]
  Day 80 | 77.0 [60.4 to 87.3] | 75.3 [58.9 to 85.9]
  Day 90 | 77.0 [60.4 to 87.3] | 71.5 [54.0 to 83.3]

25. Secondary Outcome: Time to Death
Description: Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 90
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | NA [NA to NA] — Median and 95% confidence interval could not be calculated since an insufficient number of participants had an event. | NA [NA to NA] — Median and 95% confidence interval could not be calculated since an insufficient number of participants had an event.

26. Secondary Outcome: Time to Discharge From Intensive Care Unit (ICU)
Description: Time to discharge from ICU was defined, in days, as the time between informed consent date and the date of discharge from the ICU. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 730
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 41
days | 11.1 [7.1 to 14.9] | 13.0 [7.2 to 16.2]

27. Secondary Outcome: Time to Discharge From Hospital
Description: Time to discharge from hospital was defined, in days, as the time between informed consent date and the date of discharge from the hospital. Median survival time and the associated 95% confidence interval based on Kaplan-Meier estimation are reported.
Time Frame: Baseline up to Day 730
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 19.2 [14.4 to 30.0] | 18.3 [13.2 to 25.7]

28. Secondary Outcome: Length of Stay (LOS) in ICU and Hospital After Randomization
Time Frame: Baseline up to Day 730
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days
  Length of stay in ICU | 11.1 [1 to 54] | 12.3 [0 to 121]
  Length of stay in Hospital | 19.2 [1 to 70] | 19.3 [1 to 186]

29. Secondary Outcome: Number of ICU-free Days
Description: ICU-free days will be defined as the number of days during which the participant was not in ICU, starting from the randomization date, to Day 29, or day of discontinuation.
Time Frame: Baseline up to Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
days | 14.0 [0 to 26] | 5.5 [0 to 24]

30. Secondary Outcome: Change From Baseline in Sepsis-related Organ Failure Assessment (SOFA) Score During Stay at ICU
Description: The total SOFA Score is a composite of six sub scores representing the degree of dysfunction of six organ systems: Respiratory, Cardiovascular, Liver, Renal, Coagulation and Central Nervous System. Each organ system sub score ranges from 0 to 4 points. The total SOFA Score is the sum of the six-organ system sub scores. Accordingly, the total SOFA Score may range from a minimum score of 0 to a maximum score of 24. Higher scores indicate greater degree of dysfunction.
Time Frame: Baseline up to Day 29
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 40 | 42
Score on a scale
  Baseline | 7.9 (2.39) | 8.5 (3.01)
  Change at Day 29: number analyzed (Participants) | 16 | 24
  Change at Day 29 | -6.1 (3.30) | -5.7 (3.95)

31. Secondary Outcome: Number of Participants Categorized Based on the Chest X-ray Assessments Compared to Previous Chest X-ray Assessment
Description: Number of participants with chest X-ray assessment compared to the previous assessment were assessed and reported. Number of participants which showed improvement, remission, stabilization, and worsening compared to previous CXR were reported. Cumulative data is reported only for participants who were assessed from Day 8-10.
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 8-10, 14, and 29
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants
  Improvement at Day 1: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 10
  Improvement at Day 1: Compared to previous chest X-ray | 0 | 0
  Remission at Day 1: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 10
  Remission at Day 1: Compared to previous chest X-ray | 0 | 0
  Stabilization at Day 1: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 10
  Stabilization at Day 1: Compared to previous chest X-ray | 7 | 6
  Worsening at Day 1: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 10
  Worsening at Day 1: Compared to previous chest X-ray | 2 | 4
  Improvement at Day 2: Compared to previous chest X-ray: number analyzed (Participants) | 34 | 31
  Improvement at Day 2: Compared to previous chest X-ray | 9 | 6
  Remission at Day 2: Compared to previous chest X-ray: number analyzed (Participants) | 34 | 31
  Remission at Day 2: Compared to previous chest X-ray | 0 | 0
  Stabilization at Day 2: Compared to previous chest X-ray: number analyzed (Participants) | 34 | 31
  Stabilization at Day 2: Compared to previous chest X-ray | 17 | 17
  Worsening at Day 2: Compared to previous chest X-ray: number analyzed (Participants) | 34 | 31
  Worsening at Day 2: Compared to previous chest X-ray | 8 | 8
  Improvement at Day 3: Compared to previous chest X-ray: number analyzed (Participants) | 37 | 30
  Improvement at Day 3: Compared to previous chest X-ray | 19 | 8
  Remission at Day 3: Compared to previous chest X-ray: number analyzed (Participants) | 37 | 30
  Remission at Day 3: Compared to previous chest X-ray | 0 | 1
  Stabilization at Day 3: Compared to previous chest X-ray: number analyzed (Participants) | 37 | 30
  Stabilization at Day 3: Compared to previous chest X-ray | 17 | 17
  Worsening at Day 3: Compared to previous chest X-ray: number analyzed (Participants) | 37 | 30
  Worsening at Day 3: Compared to previous chest X-ray | 1 | 4
  Improvement at Day 4: Compared to previous chest X-ray: number analyzed (Participants) | 30 | 31
  Improvement at Day 4: Compared to previous chest X-ray | 14 | 8
  Remission at Day 4: Compared to previous chest X-ray: number analyzed (Participants) | 30 | 31
  Remission at Day 4: Compared to previous chest X-ray | 1 | 3
  Stabilization at Day 4: Compared to previous chest X-ray: number analyzed (Participants) | 30 | 31
  Stabilization at Day 4: Compared to previous chest X-ray | 15 | 12
  Worsening at Day 4: Compared to previous chest X-ray: number analyzed (Participants) | 30 | 31
  Worsening at Day 4: Compared to previous chest X-ray | 0 | 8
  Improvement at Day 5: Compared to previous chest X-ray: number analyzed (Participants) | 20 | 24
  Improvement at Day 5: Compared to previous chest X-ray | 5 | 8
  Remission at Day 5: Compared to previous chest X-ray: number analyzed (Participants) | 20 | 24
  Remission at Day 5: Compared to previous chest X-ray | 2 | 2
  Stabilization at Day 5: Compared to previous chest X-ray: number analyzed (Participants) | 20 | 24
  Stabilization at Day 5: Compared to previous chest X-ray | 7 | 9
  Worsening at Day 5: Compared to previous chest X-ray: number analyzed (Participants) | 20 | 24
  Worsening at Day 5: Compared to previous chest X-ray | 6 | 5
  Improvement at Day 6: Compared to previous chest X-ray: number analyzed (Participants) | 29 | 26
  Improvement at Day 6: Compared to previous chest X-ray | 11 | 12
  Remission at Day 6: Compared to previous chest X-ray: number analyzed (Participants) | 29 | 26
  Remission at Day 6: Compared to previous chest X-ray | 1 | 2
  Stabilization at Day 6: Compared to previous chest X-ray: number analyzed (Participants) | 29 | 26
  Stabilization at Day 6: Compared to previous chest X-ray | 15 | 10
  Worsening at Day 6: Compared to previous chest X-ray: number analyzed (Participants) | 29 | 26
  Worsening at Day 6: Compared to previous chest X-ray | 2 | 2
  Improvement at Day 7: Compared to previous chest X-ray: number analyzed (Participants) | 18 | 22
  Improvement at Day 7: Compared to previous chest X-ray | 8 | 8
  Remission at Day 7: Compared to previous chest X-ray: number analyzed (Participants) | 18 | 22
  Remission at Day 7: Compared to previous chest X-ray | 0 | 0
  Stabilization at Day 7: Compared to previous chest X-ray: number analyzed (Participants) | 18 | 22
  Stabilization at Day 7: Compared to previous chest X-ray | 7 | 11
  Worsening at Day 7: Compared to previous chest X-ray: number analyzed (Participants) | 18 | 22
  Worsening at Day 7: Compared to previous chest X-ray | 3 | 3
  Improvement at Days 8-10: Compared to previous chest X-ray: number analyzed (Participants) | 27 | 22
  Improvement at Days 8-10: Compared to previous chest X-ray | 8 | 9
  Remission at Days 8-10: Compared to previous chest X-ray: number analyzed (Participants) | 27 | 22
  Remission at Days 8-10: Compared to previous chest X-ray | 3 | 3
  Stabilization at Days 8-10: Compared to previous chest X-ray: number analyzed (Participants) | 27 | 22
  Stabilization at Days 8-10: Compared to previous chest X-ray | 11 | 7
  Worsening at Days 8-10: Compared to previous chest X-ray: number analyzed (Participants) | 27 | 22
  Worsening at Days 8-10: Compared to previous chest X-ray | 5 | 3
  Improvement at Day 14: Compared to previous chest X-ray: number analyzed (Participants) | 21 | 15
  Improvement at Day 14: Compared to previous chest X-ray | 10 | 10
  Remission at Day 14: Compared to previous chest X-ray: number analyzed (Participants) | 21 | 15
  Remission at Day 14: Compared to previous chest X-ray | 1 | 1
  Stabilization at Day 14: Compared to previous chest X-ray: number analyzed (Participants) | 21 | 15
  Stabilization at Day 14: Compared to previous chest X-ray | 5 | 3
  Worsening at Day 14: Compared to previous chest X-ray: number analyzed (Participants) | 21 | 15
  Worsening at Day 14: Compared to previous chest X-ray | 5 | 1
  Improvement at Day 29: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 14
  Improvement at Day 29: Compared to previous chest X-ray | 3 | 6
  Remission at Day 29: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 14
  Remission at Day 29: Compared to previous chest X-ray | 3 | 2
  Stabilization at Day 29: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 14
  Stabilization at Day 29: Compared to previous chest X-ray | 2 | 4
  Worsening at Day 29: Compared to previous chest X-ray: number analyzed (Participants) | 9 | 14
  Worsening at Day 29: Compared to previous chest X-ray | 1 | 2

32. Secondary Outcome: Change in the Ratio of the Partial Pressure of Oxygen to the Fraction of Inspired Oxygen (PaO2/FiO2 Ratio)
Time Frame: Baseline up to Day 7
Population: The safety population included all randomized participants who received at least one dose of the study treatment. Here "number analyzed" n are the participants who were evaluable for this outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: P/F ratio
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
P/F ratio
  Baseline | 131.6 (55.14) | 278.6 (981.67)
  Change at Day 7: number analyzed (Participants) | 30 | 33
  Change at Day 7 | 74.6 (97.20) | 78.4 (68.57)

33. Secondary Outcome: Number of Participants Requiring Mechanical Ventilation or Non-invasive Ventilation Twelve Hours After the Second Investigational Medicinal Product (IMP) Infusion
Time Frame: Day 3: 0 to 12 hours post-IMP infusion
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 31 | 37

34. Secondary Outcome: Number Participants Using Rescue Antibiotics
Description: Any new intravenous antibiotic for CABP indication that was started after Day 1 and before Day 29 was considered a rescue antibiotic.
Time Frame: Baseline up to Day 29
Population: The safety population included all randomized participants who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cx611 160 mL
Number analyzed (Participants) | 41 | 42
Participants | 28 | 32

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started from the signature of the informed consent (Baseline) up to Day 730
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Cx611 160 mL
All-Cause Mortality (participants affected / at risk) | 12/41 | 13/42
Serious Adverse Events (participants affected / at risk) | 20/41 | 24/42
Other Adverse Events (participants affected / at risk) | 41/41 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Cx611 160 mL (N=42)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 4 (4) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Cx611 160 mL (N=42)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 8 (8)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thymus disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 6 (6)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Primary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5)
Asthenia (General disorders) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 5 (5)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Citrobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Axillary nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Akinesia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 4 (4)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03158727/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT03158727/SAP_001.pdf